CLINICAL TRIAL: NCT04919564
Title: Low Dose Continuous Furosemide Effect on Cardiac Surgery Patients With Kidney Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cardiovascular Center Harapan Kita Hospital Indonesia (Other)
Responsible Party: Principal Investigator, Prieta Adriane MD, Principal Investigator, National Cardiovascular Center Harapan Kita Hospital Indonesia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LB.02.01/VII/533/KEP024/2021; NationalCCHK (Other: National Cardiac Center Harapan Kita)
Record Dates: First submitted 2021-05-27; First posted 2021-06-09 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-03

CONDITIONS: Chronic Kidney Disease; Cardiac Disease
Keywords: Furosemide; Kidney Dysfunction; Glomerular Filtration Rate
MeSH Terms: conditions — Renal Insufficiency, Chronic; Heart Diseases | interventions — Furosemide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Allocation group was blinded for participants, care provider, and investigators
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Furosemide group (Experimental): Continuous furosemide 2 mg/hour for a period of 12 hours begins since anesthetic induction
  Interventions: Drug: Furosemide in 0.9 % NaCl 100 Mg/100 mL (1 mg/mL)
- Placebo group (Placebo Comparator): Continuous NaCl 0.9% 2 cc/hour for a period of 12 hours begins since anesthetic induction
  Interventions: Drug: NaCl 0.9%

INTERVENTIONS:
Drug: Furosemide in 0.9 % NaCl 100 Mg/100 mL (1 mg/mL) — Furosemide 2 mg/hour infusion for 12 hours since induction
  Other Names: Lasix injection
  Arms: Furosemide group
Drug: NaCl 0.9% — NaCl 0.9% 2 cc/hour for a period of 12 hours since anesthetic induction
  Arms: Placebo group

SUMMARY:
Chronic kidney disease is an independent risk factor for cardiovascular disease associated with increased mortality rate during cardiac surgery in proportion to the kidney function. Chronic kidney disease is defined by decreased glomerular filtration rate (GFR) as classified by Kidney Disease: Improving Global Outcome (KDIGO). Deterioration of kidney function has a complex and multifactorial pathophysiologic derangement. In order to counter kidney injury associated with cardiac surgery, several pharmacologic and non-pharmacologic interventions have been studied to prevent perioperative deterioration of kidney function. Diuretics as pharmacologic measure are often used post-cardiac surgery to treat fluid overload and managing patient with acute kidney injury by preventing anuria. Loop diuretics (furosemide) may improve renal blood flow, decrease reabsorption in renal tubules, decrease oxygen demand and energy consumption (blocking potassium/sodium/2cloride co-transport in loop of Henle), and prevent hypoxic injury of renal medulla. Low dose continuous furosemide hypothetically has a protective effect on cardiac surgery patients with kidney dysfunction, measured improved glomerular filtration rate, decreased indication for therapeutic furosemide infusion, and decreased need of renal replacement therapy. On the other hand, administration of furosemide is rather harmful in severe kidney dysfunction. Therefore, the objective of this study is to determine the protective effect of low-dose continuous furosemide perioperative in cardiac surgery patients with mild to moderate kidney dysfunction.

DETAILED DESCRIPTION:
The study was a double-blind randomized controlled trial to determine the protective effect of low-dose continuous furosemide perioperative in cardiac surgery patients with mild to moderate kidney dysfunction. Ethical clearance for the study was approved by Institutional Review Board of National Cardiovascular Center Harapan Kita. Patients eligible for the study was recruited and written informed consent was obtained after clear explanation of the study. Allocation of furosemide and control group was done using simple computer randomization by staff who was not involved in the study. Furosemide infusion and normal saline was prepared by independent pharmacist blinded to the study. Furosemide solution was prepared to contain 40 mg of furosemide diluted with normal saline to a total volume of 40 cc (1 mg / 1 cc) and control solution was prepared to contain only 40 cc of normal saline. Both solution was packaged in 50-cc syringe and prepared in similar fashion. The solution was administered after induction of anesthesia with rate of 2 cc per hour for 12 hours.

Baseline participant were collected before surgery. All cardiac surgery procedure was done in concordance to hospital standard operating procedure. The primary outcomes of the study were glomerular filtration rate, need of diuretic infusion dose after intervention, need of renal replacement therapy and the secondary outcomes were ICU length of stay and in hospital mortality. The calculated sample size estimated was 41 participants per group, accounting for drop-out rate, expected sample size was 45 participants per group (90 participants in total).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years old.
* Patient planned with elective cardiac surgery such as CABG, one cardiac valve replacement, one cardiac valve repair or two valves, CABG and replacement/repair one cardiac valve.
* Cardiac surgery performed using cardiopulmonary bypass machine.
* Patient with mild to moderate kidney dysfunction (GFR 30-89 mL/min/1.73m2) and never got renal replacement therapy before.

Exclusion Criteria:

* Cardiac ejection fraction <40%.
* Patient with new preoperative acute renal failure by any cause.
* Sudden shift in cardiac surgery timing (emergency cardiac surgery or repeated procedure).
* Complex cardiac disease associated with intra aortic balloon pump use, replacement of more than two cardiac valves, coronary artery disease with severe valve disease, and patient with pulmonary hypertension, and cardiac surgery procedures for congenital heart disease.
* Patient with aortic abnormality, and/or has direct effect on renal artery.
* Patients concurrently enrolled in other study with other drugs being studied.
* Patient with hemodynamic disturbance caused by hemorrhage, sepsis, anaphylactic, or cardiogenic shock.
* Patient refuses to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bambang Widyantoro, PhD, Study Director — National Cardiovascular Center Harapan Kita
Locations (1):
- National Cardiovascular Center Harapan Kita Jakarta, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Furosemide: Low dose continuous furosemide 2 mg/hour for a period of 12 hours since anesthetic induction
  Furosemide: Furosemide 2 mg/hour for 12 hours since induction
- Control: NaCl 0.9% 2 cc/hour for a period of 12 hours since anesthetic induction
  Control: NaCl 0.9% 2 cc/hour for a period of 12 hours since anesthetic induction
Period: Overall Study
Arm/Group | Furosemide | Control
Started | 45 | 45
Completed | 43 | 44
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Furosemide | Control | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (7) | 57 (8) | 58 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 12 | 19
  Male | 38 | 33 | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 45 | 45 | 90
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kilogram] | 68.7 (10.7) | 66.7 (16) | 67.7 (13.5)
Height [Mean (Standard Deviation); unit: centimeter] | 161.6 (7.93) | 160.6 (7.4) | 161.2 (7.64)
Type of operation [Count of Participants; unit: Participants]
  CABG | 36 | 29 | 65
  Valve surgery | 8 | 16 | 24
  CABG + Valve Surgery | 1 | 0 | 1
percentage of Left Ventricular ejection fraction [Mean (Standard Deviation); unit: %] | 56.91 (9.48) | 54.93 (9.68) | 55.92 (9.58)
percentage of patient with pre-operation Comorbid [Count of Participants; unit: Participants] — Measure the Charlson Comorbidity Index (CCI) score for participant with following comorbidity; Myocardial infarction 1, Congestive heart failure 1, Peripheral vascular disease 1, Dementia 1, Chronic pulmonary disease 1, Rheumatological disease 1, Peptic ulcer disease 1, Mild liver disease 1, Diabetes without chronic complications 1, Diabetes with chronic complications 2, Hemiplegia or paraplegia 2, Renal disease 2, Solid tumor 2, Leukemia 2, Lymphoma 2, Moderate or severe liver disease 3, Human immunodeficiency virus/Acquired immunodeficiency syndrome 6, Metastatic solid tumor 6
  Participants
    score 1-2 (mild condition) | 41 | 41 | 82
    score 3-4 (moderate condition) | 3 | 4 | 7
    score >5 (severe condition) | 1 | 0 | 1
patient with history of daily use of ACEI/ARB [Count of Participants; unit: Participants]
  history of ACE-i/ARB | 30 | 32 | 62
  no history of ACE-i/ARB | 15 | 13 | 28
patient with history of daily use of Diuretic [Count of Participants; unit: Participants]
  History of Diuretics | 19 | 25 | 44
  no History of Diuretics | 26 | 20 | 46
percentage of patient with pre operation renal Dysfunction [Count of Participants; unit: Participants]
  mildly impaired | 22 | 22 | 44
  moderately impaired | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Glomerular Filtration Rate at Baseline
Description: Glomerular Filtration Rate measured at baseline
Time Frame: baseline / before induction to anesthesia
Measure: Median (Full Range); unit: mL/mnt/1.73 m^2
Arm/Group | Furosemide | Control
Number analyzed (Participants) | 45 | 45
mL/mnt/1.73 m^2 | 56 [30 to 88] | 67 [35 to 89]

2. Primary Outcome: Glomerular Filtration Rate at 12 Hours From Drug Infusion
Description: Glomerular Filtration Rate measured at 12 hours from the initiation of drug infusion
Time Frame: 12 hours from drug infusion
Measure: Median (Full Range); unit: mL/mnt/1.73 m^2
Arm/Group | Furosemide | Control
Number analyzed (Participants) | 43 | 44
mL/mnt/1.73 m^2 | 45 [14 to 84] | 46 [19 to 99]

3. Primary Outcome: Glomerular Filtration Rate at 24 Hours From Drug Infusion
Description: Glomerular Filtration Rate measured at 24 hours from the initiation of drug infusion
Time Frame: 24 hours after from infusion
Measure: Median (Full Range); unit: mL/mnt/1.73 m^2
Arm/Group | Furosemide | Control
Number analyzed (Participants) | 43 | 44
mL/mnt/1.73 m^2 | 39.5 [21 to 87] | 38 [10 to 73]

4. Primary Outcome: Glomerular Filtration Rate at 48 Hours From Drug Infusion
Description: Glomerular Filtration Rate measured at 48 hours from the initiation of drug infusion
Time Frame: 48 hours from drug infusion
Measure: Median (Full Range); unit: mL/mnt/1.73 m^2
Arm/Group | Furosemide | Control
Number analyzed (Participants) | 43 | 44
mL/mnt/1.73 m^2 | 41 [15 to 89] | 41.5 [9 to 84]

5. Primary Outcome: Glomerular Filtration Rate at 120 Hours From Drug Infusion
Description: Glomerular Filtration Rate measured at 120 hours from the initiation of drug infusion
Time Frame: 120 hours from drug infusion
Measure: Median (Full Range); unit: mL/mnt/1.73 m^2
Arm/Group | Furosemide | Control
Number analyzed (Participants) | 43 | 44
mL/mnt/1.73 m^2 | 49 [22 to 103] | 50 [15 to 98]

6. Primary Outcome: Therapeutic Dose of Continuous Diuretic Infusion
Description: number of participants with Therapeutic Dose of Continuous Diuretic Infusion
Time Frame: 28 days (or until hospital discharge)
Measure: Count of Participants; unit: Participants
Arm/Group | Furosemide | Control
Number analyzed (Participants) | 43 | 44
Participants | 10 | 23

7. Primary Outcome: Renal Replacement Therapy
Description: number of participant with Renal Replacement Therapy
Time Frame: 28 days (or until hospital discharge)
Measure: Count of Participants; unit: Participants
Arm/Group | Furosemide | Control
Number analyzed (Participants) | 43 | 44
Participants | 4 | 1

8. Secondary Outcome: ICU Length of Stay
Description: The length of stay in ICU
Time Frame: 28 days (or until hospital discharge)
Measure: Median (Full Range); unit: hours
Arm/Group | Furosemide | Control
Number analyzed (Participants) | 43 | 44
hours | 27 [13 to 340] | 24 [9 to 384]

9. Secondary Outcome: In Hospital Mortality
Description: number of In Hospital mortality
Time Frame: 28 days (or until hospital discharge)
Measure: Count of Participants; unit: Participants
Arm/Group | Furosemide | Control
Number analyzed (Participants) | 43 | 44
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: 30 days since administration of Furosemide or control
Description: adverse event are to be reported:
  1. All-Cause Mortality: The occurrence of death due to any cause
  2. Serious Adverse event adverse event expected: hypovolemia , negative fluid balance more than -2000mL/24 hours, Na<135 mEq/L, acid imbalance, Sign of acute hearing loss
Arm/Group | Furosemide | Control
All-Cause Mortality (participants affected / at risk) | 1/43 | 1/44
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/44
Other Adverse Events (participants affected / at risk) | 0/43 | 0/44

LIMITATIONS AND CAVEATS:
Technical problems with measurement leading to unreliable or uninterpretable data; others attendings decision leading to termination of subject

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-24): https://cdn.clinicaltrials.gov/large-docs/64/NCT04919564/Prot_SAP_000.pdf